CLINICAL TRIAL: NCT01994278
Title: Comparison of Soft Toothbrush and Brushless Cleaner in Their Ability to Remove Plaque From Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peri-Swab, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 12-038A
Record Dates: First submitted 2012-07-31; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-04

CONDITIONS: Plaque Control

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tooth brush (Experimental): Periclean is a soft rubber gentle toothbrush
  Interventions: Device: Peri Clean

INTERVENTIONS:
Device: Peri Clean

SUMMARY:
The aim of this study is to observe whether a brushless cleaning device can be equally as effective in removing plaque from the teeth as a soft toothbrush. The goal is to give people an alternative to bristle brush cleaning if they find they are brushing too hard. The hypothesis is that it is possible to maintain healthy teeth and gingiva by using brushless methods in conjunction with flossing.

ELIGIBILITY:
Inclusion Criteria:

* 18 yrs of age
* healthy gingiva

Exclusion Criteria:

* less than 18 yrs old
* patients with braces
* decisionally impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Silness Gingival index | June 2013
  using a periodontal probe gently between the tooth and gum